CLINICAL TRIAL: NCT02223702
Title: Clinical Evaluation of Systemic Moxifloxacin Compared to Amoxicillin Plus Metronidazole Adjunct to Non-surgical Treatment in Generalized Aggressive Periodontitis: A Randomized Clinical Trial
Brief Title: Alternative Antibiotic Regime in the Treatment of GAgP
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Kocaeli University (Other)
Responsible Party: Principal Investigator, Esra Guzeldemir-Akcakanat, Associate Professor, Kocaeli University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: KOUKAEK5/9
Record Dates: First submitted 2014-08-20; First posted 2014-08-22 (Estimated); Results first posted 2018-11-02 (Actual); Last update posted 2018-11-02 (Actual); Status verified 2018-02

CONDITIONS: Generalized Aggressive Periodontitis; Aggressive Periodontitis
Keywords: Aggressive periodontitis; amoxicillin; metronidazole; moxifloxacin; nonsurgical periodontal debridement.
MeSH Terms: conditions — Aggressive Periodontitis | interventions — Amoxicillin; Metronidazole; Moxifloxacin

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- amoxicillin+metronidazole (Active Comparator): amoxicillin+metronidazole group received a combination of 500 mg of amoxicillin and 500 mg metronidazole three times per day for 7 days.
  Interventions: Drug: Amoxicillin; Drug: Metronidazole
- moxifloxacin (Experimental): The moxifloxacin group received 400 mg moxifloxacin, once in a day for 7 days.
  Interventions: Drug: Moxifloxacin

INTERVENTIONS:
Drug: Amoxicillin — 500 mg, 3 times per day for 7 days
  Other Names: largopen
  Arms: amoxicillin+metronidazole
Drug: Metronidazole — 500 mg, 3 times per day, for 7 days
  Other Names: flagyl
  Arms: amoxicillin+metronidazole
Drug: Moxifloxacin — 400 mg, once in a day for 7 days.
  Other Names: pitoxil
  Arms: moxifloxacin

SUMMARY:
The objective of this randomized clinical study was to evaluate the effect of systemic administration of moxifloxacin compared to amoxicillin plus metronidazole combined with non-surgical treatment in patients with generalized aggressive periodontitis (GAgP) in 6-month follow-up.

A total of 40 systemically healthy patients with GAgP will evaluate in this randomized clinical trial. Periodontal parameters (plaque index, gingival index, probing depth, bleeding on probing, clinical attachment level) will be recorded at baseline, 1st, 3rd and 6th month. Patients will receive either 400 mg moxifloxacin per os once daily or 500 mg metronidazole and 500 mg amoxicillin per os three times daily for 7 days consecutively.

DETAILED DESCRIPTION:
The American Academy of Periodontology and the European Federation of Periodontology were reported that patients with GAgP may have benefit from adjunctive administration of antibiotics. Antibiotics are used as an adjunct to nonsurgical treatment either locally or systemically. Systemic antimicrobial agents as adjunct to nonsurgical treatment provide additional benefits over mechanical therapy alone in terms of probing depth reduction and periodontal attachment gain.

Amoxicillin is a moderate spectrum, bacteriolytic β-lactam antibiotic, and metronidazole which is active against anaerobic bacteria is a nitroimidazole. scaling and root planing combination with metronidazole plus amoxicillin therapy was found to be more effective in suppressing P. gingivalis and eradication of A. actinomycetemcomitans and preventing re-colonization of A. actinomycetemcomitans because of the synergistic effect of this combination and their wide spectrum of activity. It was found to be superior to azithromycin, doxycycline, and metronidazole in the treatment of GAgP.

Quinolones were introduced for use in urinary tract infections in the 1970s. Moxiflocaxin is a fourth generation fluoroquinolone antibiotic exhibits good tissue penetration and high oral bioavailability and has improved activity against Gram- positive, aerobic and anaerobes. Moxifloxacin is used in the systemic treatment of respiratory infections, acute sinusitis, odontogenic abscesses, osteomyelitis of the mandible and locally in the treatment of ophthalmic infections.

Moxiflocaxin has good activity against putative periodontal pathogens, including Porphyromonas gingivalis, Tanneralla forsythia, Prevotella spp, Fusobacterium nucleatum, Actinomyces spp, Campylobacter rectus, Peptostreptococcus spp. and Aggregatibacter actinomycetemcomitans, located within biofilm or intracellulary. It was shown that A.a. strains were highly susceptible to fluoro-quinolones ciprofloxacin and moxifloxacin. Some of the adjunctive antibiotics are secreted in saliva in insufficient concentrations to inhibit A.a. Moxifloxacin seems to be secreted in saliva at higher levels than in plasma and may also concentrate at the site of infection since it penetrates polymorphonuclear granulocytes and epithelial cells. Moxifloxacin was found to be superior to clindamycin, metronidazole or doxycycline.

Systemic administration of moxifloxacin as an adjunct to scaling and root planing was found to be more effective compared to scaling and root planing alone or scaling and root planing in conjunction with doxycycline in the treatment of severe chronic periodontitis. To best our knowledge, there is no study that evaluates the effect of moxifloxacin adjunct to scaling and root planing in the treatment of GAgP.

The aim of this single center, randomized clinical study was to evaluate the impact of adjunctive systemic moxifloxacin compared to the use of adjunctive systemic amoxicillin and metronidazole during full-mouth scaling and root planing on the success of the treatment of patients with GAgP with 6-month follow-up. The hypothesis was the use of adjunctive systemic moxifloxacin would provide the similar clinical results as adjunct systemic amoxicillin and metronidazole during scaling and root planing.

This study was a single-center, randomized, parallel-design clinical trial with 6 month follow-up. It was conducted at Kocaeli University, Faculty of Dentistry, Department of Periodontology between 2011-2013. The study protocol was approved by the Ethics Committee of the Medical Faculty of Kocaeli University (KOU KAEK 5/9) and was conducted in accordance with the Helsinki declaration of 1975, as revised in 2000.

The GAgP patients were recruited from patients seeking periodontal treatment at Kocaeli University, Faculty of Dentistry, Department of Periodontology, Kocaeli, Turkey. Approximately, 12.000 patients were screened the dates between June 2011 and September 2012. A complete medical, dental, periodontal and radiographic examination was performed. The study protocol explained to the patients. From patients who willing to participate to the study, written informed consent was obtained and included the study.

The periodontal diagnosis of subjects with GAgP was established on the basis of clinical and radiographic criteria defined by the 1999 International World Workshop for a Classification of Periodontal Diseases and Conditions. Patients were included if they were between 18 and 35 years of age and otherwise healthy. The bone loss estimation was radiographically performed in each patient for the assessment of the extent and severity of alveolar bone loss. Medical and dental histories were questioned. Subjects were excluded if they had any known systemic diseases or conditions that can/could influence the periodontal status (cancer, cardiovascular and respiratory diseases), history of hepatitis or HIV infection, immunosuppressive chemotherapy, current pregnancy, planning a pregnancy or lactation, requirement for antibiotic prophylaxis, oral diseases other than GAgP, ongoing orthodontic therapy, a history of antibiotic therapy or periodontal treatment within the preceding six months. Subjects were excluded if they had known allergies to quinolones or penicillin or metronidazole.

Periodontal Examination The full-mouth clinical periodontal measurements were recorded at 6 sites per tooth (mesio-buccal, mid-buccal, disto-buccal, disto-lingual, mid-lingual, and mesio-lingual) including plaque index (PI), gingival index (GI), probing depth (PD), bleeding on probing (BOP) and clinical attachment level (CAL). CAL was calculated from the cement-enamel junction to the base of the periodontal pocket. Williams periodontal probe was used for periodontal measurements. All measurements and scaling and root planing were performed by the same single calibrated and trained periodontist in a standardized manner.

Allocation concealment The patients were randomly assigned to one of the study groups. To ensure complete masking of allocation, before the recruitment of the patients, forty identical, opaque-colored, impermeable plastic bags which include toothbrush, interproximal brush, toothpaste and either moxifloxacin or amoxicillin and metronidazole were prepared and coded. A code number was given to each subject. Randomization codes were kept separately from the clinical evaluation forms by one of the authors until the treatment and follow-up visits were completed. The examiner who performed the treatment was unaware of the allocation.

Prior to treatment, all subjects were gone through motivation sessions for oral hygiene.

Following to periodontal measurements, full-mouth supragingival scaling using ultrasonic scaler and polishing were performed, and a toothbrush, toothpaste and an interproximal toothbrush were provided to all subjects. One week later, the patients were examined for plaque accumulation and oral hygiene. The patients who cannot maintain proper oral hygiene were excluded from the study. Only 39 patients fulfilled the qualification criteria for enrollment for the present study.

Subjects were randomly assigned to receive one of the two treatment groups. Moxifloxacin group received scaling and root planing and an adjunctive systemic antibiotic, 400 mg moxifloxacin, once in a day for 7 days and amoxicillin and metronidazole group received a combination of 500 mg of amoxicillin and 500 mg metronidazole three times per day for 7 days. The subjects were instructed to take first dose of the antibiotics in the morning of the first session since the microorganisms are organized on the root surface and protected from antimicrobial agents. Scaling and root planing were performed on 2 consecutive days in 24 hours under the local anesthesia. On each day, scaling and root planing were performed in 2 quadrants using ultrasonic scalers and manual instruments . The endpoint of scaling and root planing was a tactile smooth root surface.

The subjects were insistently informed about the intake of the antibiotics properly, and they asked to inform the researches if they needed to take another antibiotics or anti-inflammatory agents for another reason during and following the study for 6 months.

Patients used a 0.2% chlorhexidine digluconate rinse twice a day for a month and brushed their teeth by tooth brushes and interproximal tooth brushes twice a day. Patients asked to report any adverse events and side effects of the antimicrobial agents as soon as possible.

Subjects were monitored one week after the second scaling and root planing session. At this session, antibiotic intake, adverse events and side effects were questioned; oral hygiene and plaque accumulation were controlled. Subjects were screened at 1, 3 and 6 months after completion of nonsurgical treatment. During these sessions, clinical periodontal parameters, any medical history change, especially, whether antibiotic therapy had been prescribed for any reason was recorded. At the end of these sessions, supragingival scaling was performed, if needed.

The present study was conducted within in the same clinic, and the patients were taken to the same dental chair and treated with a same experienced periodontist for to discard discrepancies and to provide standardized and controlled environment.

Sample size calculation

The primary outcome variable was probing depth changes. The sample size was calculated based on previous information from a study conducted in our department, using data relative to the mean difference and standard deviation (SD) between the experimental periods for the probing depth parameters.57 Considering a mean probing depth difference of 1.3 mm between evaluation periods, it was estimated that 13 patients for each group would be necessary to provide 95% power (0.54 SD, α error of 0.05, and β error of 0.2).58 However, we aimed to recruit 20 patients to each group if we lose to follow the patients during the study.

ELIGIBILITY:
Inclusion Criteria:

* The periodontal diagnosis of subjects with GAgP was established on the basis of clinical and radiographic criteria defined by the 1999 International World Workshop for a Classification of Periodontal Diseases and Conditions.
* Patients were included if they were between 18 and 35 years of age and otherwise healthy.

Exclusion Criteria:

* if the patients had any known systemic diseases or conditions that can/could influence the periodontal status (cancer, cardiovascular and respiratory diseases)
* history of hepatitis or HIV infection,
* immunosuppressive chemotherapy
* current pregnancy, planning a pregnancy or lactation
* requirement for antibiotic prophylaxis
* oral diseases other than GAgP, ongoing orthodontic therapy
* a history of antibiotic therapy or periodontal treatment within the preceding six months.
* Subjects were excluded if they had known allergies to quinolones or penicillin or metronidazole
* Not willing to participate to the study.
* Not accept to sign written informed consent

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 39 (Actual)
Dates: Start 2011-05; Primary Completion 2012-05 (Actual); Study Completion 2014-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Esra Guzeldemir-Akcakanat, Principal Investigator — Kocaeli University
Locations (1):
- Kocaeli University Faculty of Dentistry Department of Periodontology, Kocaeli, Turkey (Türkiye)

REFERENCES:
- [Background] Guentsch A, Jentsch H, Pfister W, Hoffmann T, Eick S. Moxifloxacin as an adjunctive antibiotic in the treatment of severe chronic periodontitis. J Periodontol. 2008 Oct;79(10):1894-903. doi: 10.1902/jop.2008.070493. PMID 18834244
- [Background] Sobottka I, Cachovan G, Sturenburg E, Ahlers MO, Laufs R, Platzer U, Mack D. In vitro activity of moxifloxacin against bacteria isolated from odontogenic abscesses. Antimicrob Agents Chemother. 2002 Dec;46(12):4019-21. doi: 10.1128/AAC.46.12.4019-4021.2002. PMID 12435716
- [Result] Herrera D, Sanz M, Jepsen S, Needleman I, Roldan S. A systematic review on the effect of systemic antimicrobials as an adjunct to scaling and root planing in periodontitis patients. J Clin Periodontol. 2002;29 Suppl 3:136-59; discussion 160-2. doi: 10.1034/j.1600-051x.29.s3.8.x. PMID 12787214
- [Result] Mestnik MJ, Feres M, Figueiredo LC, Duarte PM, Lira EA, Faveri M. Short-term benefits of the adjunctive use of metronidazole plus amoxicillin in the microbial profile and in the clinical parameters of subjects with generalized aggressive periodontitis. J Clin Periodontol. 2010 Apr;37(4):353-65. doi: 10.1111/j.1600-051X.2010.01538.x. PMID 20447259
- [Result] Sgolastra F, Petrucci A, Gatto R, Monaco A. Effectiveness of systemic amoxicillin/metronidazole as an adjunctive therapy to full-mouth scaling and root planing in the treatment of aggressive periodontitis: a systematic review and meta-analysis. J Periodontol. 2012 Jun;83(6):731-43. doi: 10.1902/jop.2011.110432. Epub 2011 Nov 3. PMID 22050545
- [Result] Herrera D, Alonso B, Leon R, Roldan S, Sanz M. Antimicrobial therapy in periodontitis: the use of systemic antimicrobials against the subgingival biofilm. J Clin Periodontol. 2008 Sep;35(8 Suppl):45-66. doi: 10.1111/j.1600-051X.2008.01260.x. PMID 18724841
- [Result] Xajigeorgiou C, Sakellari D, Slini T, Baka A, Konstantinidis A. Clinical and microbiological effects of different antimicrobials on generalized aggressive periodontitis. J Clin Periodontol. 2006 Apr;33(4):254-64. doi: 10.1111/j.1600-051X.2006.00905.x. PMID 16553634
- [Derived] Khattri S, Kumbargere Nagraj S, Arora A, Eachempati P, Kusum CK, Bhat KG, Johnson TM, Lodi G. Adjunctive systemic antimicrobials for the non-surgical treatment of periodontitis. Cochrane Database Syst Rev. 2020 Nov 16;11(11):CD012568. doi: 10.1002/14651858.CD012568.pub2. PMID 33197289

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Amoxicillin+Metronidazole | Moxifloxacin
Started | 20 | 19
Completed | 19 | 15
Not Completed | 1 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Amoxicillin+Metronidazole | Moxifloxacin | Total
Number analyzed (Participants) | 20 | 19 | 39
Age, Customized [Number; unit: participants]
  years (older than 18 years, younger than 35 years) | 20 | 19 | 39
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 9 | 19
  Male | 10 | 10 | 20
Region of Enrollment [Number; unit: participants]
  Turkey | 20 | 19 | 39

OUTCOME MEASURES:

1. Primary Outcome: The Primary Outcome Variable Was Probing Depth.
Description: We measured the probing depth at baseline, 1st, 3rd and 6th months. The changes were evaluated among and between groups.
Time Frame: 6-months
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Amoxicillin+Metronidazole | Moxifloxacin
Number analyzed (Participants) | 19 | 15
mm
  Baseline | 4.57 (1.08) | 4.18 (0.62)
  1st month | 3.12 (0.68) | 2.91 (0.38)
  3rd month | 3.11 (0.6) | 2.79 (0.33)
  6th month | 3.15 (0.67) | 3.01 (0.46)
Statistical Analysis 1: Comparison: Amoxicillin+Metronidazole vs Moxifloxacin; Test type: Superiority or Other; p < 0.01, Friedman Test; All rows were compared to eachother

2. Secondary Outcome: The Attachment Loss Were Considered as a Secondary Measure.
Description: Attachment loss were recorded at baseline, 1st, 3rd and 6th months as millimeters. The data were compared among and between groups.
Time Frame: 6-months
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Amoxicillin+Metronidazole | Moxifloxacin
Number analyzed (Participants) | 20 | 19
mm
  Baseline | 5.03 (1.14) | 4.94 (0.81)
  1st month | 4.37 (0.87) | 4.14 (0.87)
  3rd month | 4.41 (0.93) | 3.98 (0.82)
  6th month | 4.33 (0.94) | 4.30 (0.93)
Statistical Analysis 1: Comparison: Amoxicillin+Metronidazole vs Moxifloxacin; Test type: Superiority or Other; p < 0.01, ANOVA; All rows were compared to eachother

ADVERSE EVENTS:
Arm/Group | Amoxicillin+Metronidazole | Moxifloxacin
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/19
Other Adverse Events (participants affected / at risk) | 0/20 | 0/19

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes